CLINICAL TRIAL: NCT04802070
Title: A Phase I Study of Adoptive Immunotherapy With Cytokine-Induced Killer Cells in Relapsed and Non-resectable Sarcomas After Multimodal Treatment.
Brief Title: Study of Adoptive Immunotherapy in Relapsed and Non-resectable Sarcomas After Multimodal Treatment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Franca Fagioli (Other)
Responsible Party: Sponsor-Investigator, Prof. Franca Fagioli, Professor, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Organization: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.A.S.T.
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIK (Experimental)
  Interventions: Drug: Autologous CIK

INTERVENTIONS:
Drug: Autologous CIK — Lymphocytapheresis of the autologous ex-vivo CIK cell expanded in the Cell factory (4 dose levels)

SUMMARY:
Monocentric, phase I study for advanced sarcoma with adoptive immunotherapy with Cytokine-Induced Killer (CIK).

In the first part of the study Patient's' peripheral blood will be collected and CIK cell expansion and storage will occur at the Regina Margherita Children's Hospital Cell Factory.

In the second part of the study the Maximum Tolerated Dose (MTD) will be determined in order to find the Recommended Dose for Phase II (RP2D)

ELIGIBILITY:
Inclusion Criteria for part 1

* Patients with histologically documented unresectable sarcomas which progressed after first or further line treatments for relapsing disease who could be enrolled in Part 2 of study immediately or after a new line of treatment;
* Karnofsky score ≥ 70% (patients with Karnofsky score ≥ 50% are eligible if it depends solely on orthopedic problems)
* Estimated life expectancy > 3 months;
* Adequate bone marrow functions:
* Signed informed consent;
* Negative serum or urine pregnancy test within 48 hours from collection of peripheral blood or from lympho cyto apheresis (if post-pubertal female patients);
* Archived histological tumour sample available

Inclusion Criteria for part 2

* Patients with histologically documented unresectable sarcomas which progressed after a first or further line treatments for relapsing disease
* Measurable disease (bone lesions are included);
* Karnofsky score ≥ 70% (patients with Karnofsky score ≥ 50% are eligible if its depend solely on orthopedic problems)
* Estimated life expectancy > 3 months;
* Adequate bone marrow, hepatic and renal functionality
* Signed informed consent;
* Archived histological tumour sample available;
* Patients should have a venous central access;
* Pregnancy test should be negative 48 hours before treatment for post-pubertal women patients. All post-pubertal patients are to take adequate anti-contraceptive measures during treatment and until 8 weeks after the last dose of treatment.

Exclusion Criteria for part 1

* History of Human Immunodeficiency Virus, Hepatitis C Virus, Hepatitis B Virus or Hepatitis A Virus infection;
* Patients receiving chemotherapy and/or immunotherapy and/or anti-tumour agents and/or radiotherapy on more than 10% of bone marrow area two weeks before peripheral blood collection or lymphocytapheresis;
* Patients with neuro-psychiatric disorders or social or geographic problems that would prohibit the understanding or rendering informed consent and compliance with the requirements of this protocol are excluded.

Exclusion Criteria for part 2

* Patients with Ewing/Primitive Neuroectodermal Tumor Sarcoma, Rhabdomyosarcoma as well as other rapidly growing sarcomas are not to be included in the study;
* Presence of Central Nervous System metastases and/or meningeal neoplastic involvement;
* Patients with seizure disorders;
* Severe renal, vascular, cardiac, hepatic, lung disorders;
* Patients with any severe and/or uncontrolled medical conditions such as unstable angina pectoris, heart failure ≥ grade 2, a recent heart attack within 6 months, uncontrolled heart non arrhythmia uncontrolled metabolic disorders, cirrhosis, uncontrolled hypertension
* Patients with a non-optimal ex-vivo expansion of autologous CIK cells during Part 1 (< 0.5 x 107/kg CIK cells);
* History of Human Immunodeficiency Virus, Hepatitis C Virus, Hepatitis B Virus or Hepatitis A Virus infection;
* Presence of bleeding disorders;
* Patients undergoing renal dialysis;
* Presence of uncontrolled diabetes
* Patients unable to swallow oral medications;
* Patients receiving concomitant steroid or immunotherapy (except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg for adrenal insufficiency).
* Anticancer chemotherapy or experimental drugs or immunotherapy or radiotherapy 2 weeks before entering the study;
* Anticancer chemotherapy or experimental drugs or immunotherapy or radiotherapy on target lesions 2 weeks before entering the study;
* Prior exposure to CIK cells;
* Major surgery 4 weeks before entering the study;
* Minor surgery 1 week before entering the study;
* Patients with allergic reactions or hypersensibility to excipient
* Pregnant or breast-feeding patients;
* Patients with neuro-psychiatric disorders or social or geographic problems that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol are excluded.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
DLT | 6 weeks
  Incidence of dose-limiting toxicity (DLT) associated with CIK autologous cells administration

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided